CLINICAL TRIAL: NCT00702546
Title: Follow-up Protocol to Collect the Outcome of Frozen-thawed Embryo Transfer Cycles After Cryopreservation of Embryos in Clinical Trial 107012
Brief Title: Follow-up Protocol on the Outcome of Frozen-thawed Embryo Transfer Cycles From Clinical Trial P05690 (P05711)
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: P05711; 2006-003813-42 (EudraCT Number); 107015 (Other: Organon); MK-8962-004 (Other: Merck)
Record Dates: First submitted 2008-06-18; First posted 2008-06-20 (Estimated); Results first posted 2015-05-05 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: In Vitro Fertilization
Keywords: In-vitro fertilization; Controlled Ovarian Stimulation; Cumulative pregnancy data; Follow-up
MeSH Terms: interventions — follicle stimulating hormone, human, with HCG C-terminal peptide; follitropin alfa; Gonadotropin-Releasing Hormone; Progesterone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Corifollitropin alfa 100 μg: In follow-up study, no medication or investigational product was administered. But in base study P05690 (NCT00702845), participants received single subcutaneous (SC) injection of corifollitropin alfa 100 μg (Org 36286) on Day 2 or 3 of the menstrual cycle and daily placebo-recombinant Follicle Stimulating Hormone (recFSH) injections (7 total) from Stimulation Day 1 up to and including Stimulation Day 7. Participants in base study P05690 also received open-label recFSH (up to 200 IU/day) from Stimulation Day 8 onwards, up to and including Day of Human Chorion Gonadotropin (hCG) administration. Participants also received Gonadotropin Releasing Hormone (GnRH) antagonist ganirelix (0.25 mg) once daily SC starting on Stimulation Day 5 up to and including the Day of hCG (10,000 or 5,000 IU/USP). Participants also received progesterone (at least 600 mg/day vaginally or 50 mg/day IM), starting on day of oocyte pick-up (OPU) and continuing for at least 6 weeks or up to menses.
  Interventions: Drug: corifollitropin alfa; Drug: gonadatropin releasing hormone (GnRH) antagonist ganirelix; Drug: human chorion gonadatropin (hCG); Biological: progesterone; Drug: placebo-recFSH (follitropin alfa); Biological: open-label recFSH
- recFSH 150 IU: In this follow-up study, no medication or investigational product was administered. However, in base study P05690 (NCT00702845), participants in the reference group received a single SC injection of placebo-corifollitropin alfa administered on Day 2 or 3 of the menstrual cycle and daily SC recFSH 150 IU injections (7 total) from Stimulation Day 1 up to and including Stimulation Day 7. Participants also received open-label recFSH (up to 200 IU/day) from Stimulation Day 8 onwards, up to and including the day of hCG (10,000 or 5,000 IU/USP) administration. Participants also received the GnRH antagonist ganirelix (0.25 mg) once daily SC starting on Stimulation Day 5 up to and including the Day of hCG. Participants also received progesterone (at least 600 mg/day vaginally or 50 mg/day IM), starting on the day of OPU and continuing for at least 6 weeks or up to menses.
  Interventions: Biological: recFSH (follitropin alfa); Drug: gonadatropin releasing hormone (GnRH) antagonist ganirelix; Drug: human chorion gonadatropin (hCG); Biological: progesterone; Drug: placebo-corifollitropin alfa; Biological: open-label recFSH

INTERVENTIONS:
Drug: corifollitropin alfa — Single injection of 100 μg corifollitropin alfa administered under protocol P05690
  Other Names: Org 36286
  Groups: Corifollitropin alfa 100 μg
Biological: recFSH (follitropin alfa) — Daily recFSH administered under protocol P05690
  Other Names: Puregon®/Follistim®
  Groups: recFSH 150 IU
Drug: gonadatropin releasing hormone (GnRH) antagonist ganirelix — GnRH antagonist ganirelix administered SC at a dose of 0.25 mg/day under protocol P05690
Drug: human chorion gonadatropin (hCG) — hCG 5,000 IU or 10,000 IU administered SC under protocol P05690
Biological: progesterone — Under protocol P05690, progesterone was started on the day of oocyte pick-up (OPU) and continued for at least 6 weeks or up to menses. Participants received at least 600 mg/day vaginally or 50 mg/day IM.
Drug: placebo-recFSH (follitropin alfa) — Placebo-recFSH at the equivalent volume of 150 IU/day administered under protocol P05690
  Groups: Corifollitropin alfa 100 μg
Drug: placebo-corifollitropin alfa — Single SC injection of placebo-corifollitropin alfa on Day 2 or 3 of the menstrual cycle, administered under protocol P05690
  Groups: recFSH 150 IU
Biological: open-label recFSH — Open-label recFSH up to a maximum dose of 200 IU/day, administered under protocol P0590

SUMMARY:
Clinical trial objective is to collect the outcome of Frozen-Thawed Embryo Transfer (FTET) cycles performed after the embryos are cryopreserved in the base study P05690 in order to estimate the cumulative pregnancy rate for each treatment group.

DETAILED DESCRIPTION:
This is a follow-up protocol to collect the outcome of FTET cycles, performed after the embryos are cryopreserved in base study P05690 (NCT00702845), to enable estimation of the cumulative pregnancy rate for each treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Participants from whom embryos have been cryopreserved in base study P05690, of which at least one embryo is thawed for use in a subsequent FTET cycle;
* Able and willing to give written informed consent.

Exclusion Criteria:

* None

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women from whom embryos have been cryopreserved in base study P05690
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2006-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Period one consists of participants from the base study P05690 (NCT00702845) randomized to treatment groups corifollitropin alfa (Org 36286) or recombinant Follicle Stimulating Hormone (recFSH). Period two consists of eligible participants (N = 102) from the base study who enrolled in the follow up study P05711.
Groups:
- Corifollitropin Alfa 100 μg: Participants in base study P05690 received single subcutaneous (SC) injection of corifollitropin alfa 100 μg (Org 36286) on Day 2 or 3 of menstrual cycle and daily placebo-recombinant Follicle Stimulating Hormone (recFSH) injections (7 total) from Stimulation Day 1 up to and including Stimulation Day 7. Participants received open-label recFSH (up to 200 IU/day) from Stimulation Day 8 onwards, up to and including Day of Human Chorion Gonadotropin (hCG) administration. Participants also received Gonadotropin Releasing Hormone (GnRH) antagonist ganirelix (0.25 mg) once daily SC starting on Stimulation Day 5 up to and including Day of hCG (10,000 or 5,000 IU/USP); and progesterone (at least 600 mg/day vaginally or 50 mg/day IM), starting on day of oocyte pick-up (OPU) and continuing at least 6 weeks or up to menses. Eligible participants from base study were enrolled in follow up study P05711, but no study treatments were given, and embryos obtained in base study underwent FTET cycles.
- recFSH 150 IU: Participants in the reference group in base study P05690 received a single SC injection of placebo-corifollitropin alfa administered on Day 2 or 3 of the menstrual cycle and daily SC recFSH 150 IU injections (7 total) from Stimulation Day 1 up to and including Stimulation Day 7. Participants also received open-label recFSH (up to 200 IU/day) from Stimulation Day 8 onwards, up to and including the Day of hCG administration. Participants also received the GnRH antagonist ganirelix (0.25 mg) once daily SC starting on Stimulation Day 5 up to and including the Day of hCG (10,000 or 5,000 IU/USP). Participants also received progesterone (at least 600 mg/day vaginally or 50 mg/day IM), starting on the Day of OPU and continuing for at least 6 weeks or up to menses. Eligible participants from the base study were enrolled in follow up study P05711, but no study treatments were given, and embryos obtained in the base study underwent FTET cycles.
Period: Base Study P05690 (NCT00702845)
Arm/Group | Corifollitropin Alfa 100 μg | recFSH 150 IU
Started | 268 | 128
Completed | 246 (To complete study, participants from the base study P05690 (NCT00702845) had embryos transferred.) | 121 (To complete study, participants from the base study P05690 (NCT00702845) had embryos transferred.)
Not Completed | 22 | 7
Period: Follow Up Study P05711 (NCT00702546)
Arm/Group | Corifollitropin Alfa 100 μg | recFSH 150 IU
Started | 77 (Participants from base study P05690 with at least one embryo thawed for use in FTET cycle.) | 25 (Participants from base study P05690 with at least one embryo thawed for use in FTET cycle.)
Completed | 72 (Participants with embryo transfer in any FTET cycle) | 24 (Participants with embryo transfer in any FTET cycle)
Not Completed | 5 | 1

BASELINE CHARACTERISTICS:
Population: Eligible participants from base study P05690 (NCT00702845) who enrolled in follow up study P05711
Groups:
- Corifollitropin Alfa 100 μg: Participants in base study P05690 received single SC injection of corifollitropin alfa 100 μg (Org 36286) on Day 2 or 3 of menstrual cycle and daily placebo-recFSH injections (7 total) from Stimulation Day 1 up to and including Stimulation Day 7. Participants received open-label recFSH (up to 200 IU/day) from Stimulation Day 8 onwards, up to and including Day of hCG administration. Participants also received GnRH antagonist ganirelix (0.25 mg) once daily SC starting on Stimulation Day 5 up to and including Day of hCG (10,000 or 5,000 IU/USP); and progesterone (at least 600 mg/day vaginally or 50 mg/day IM), starting on Day of OPU and continuing at least 6 weeks or up to menses. Eligible participants from base study were enrolled in follow up study P05711, but no study treatments were given, and embryos obtained in base study underwent FTET cycles.
- Total: Total of all reporting groups
Arm/Group | Corifollitropin Alfa 100 μg | recFSH 150 IU | Total
Number analyzed (Participants) | 77 | 25 | 102
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.2 (3.0) | 31.2 (2.8) | 31.2 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 25 | 102
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Ongoing Pregnancy (Cumulative Ongoing Pregnancy Rate)
Description: Cumulative ongoing pregnancy rate was defined as 100 times the number of participants with an ongoing pregnancy either immediately after embryo transfer in base study P05690 (NCT00702845) or after one or more FTET cycles in follow up study P05711 following cryopreservation, divided by the total number of subjects that started treatment in base study P05690.
Time Frame: Up to 1 year after embryo transfer in base trial P05690 (NCT00702845), and FTET cycles in follow up study P05711
Population: Intent-to-Treat (ITT) group from base study P05690 (NCT00702845), which consisted of randomized participants who were treated with corifollitropin alfa or recFSH.
Measure: Number; unit: Percentage of participants
Arm/Group | Corifollitropin Alfa 100 μg | recFSH 150 IU
Number analyzed (Participants) | 268 | 128
Percentage of participants | 32.1 | 41.4
Statistical Analysis 1: Comparison: Corifollitropin Alfa 100 μg vs recFSH 150 IU; Treatment groups were compared with a generalized linear model for the cumulative ongoing pregnancy rate including covariates treatment group, age class (< 32 yrs vs. ≥ 32 yrs), planned IVF treatment (IVF vs. ICSI) and region (Europe vs. Asia); Test type: Superiority or Other; Risk Difference (RD) = -9.4, 95% CI 2-sided [-19.5 to 0.7]

2. Secondary Outcome: Percentage of Participants in Follow up Study With a Miscarriage Per Clinical Pregnancy
Description: Miscarriages were calculated per clinical pregnancy, defined as the presence of at least one gestational sac as assessed by USS or Doppler, or confirmed by live birth.
Time Frame: After one or more FTET cycles, assessed at least 10 weeks after embryo transfer (up to 1 year)
Population: Participants in follow up study P05711 with a clinical pregnancy
Measure: Number; unit: Percentage of participants
Arm/Group | Corifollitropin Alfa 100 μg | recFSH 150 IU
Number analyzed (Participants) | 22 | 10
Percentage of participants | 13.6 | 10.0

3. Secondary Outcome: Percentage of Participants in Follow up Study With a Miscarriage Per Vital Pregnancy
Description: Miscarriages were calculated per vital pregnancy, defined as the presence of at least one fetus with heart activity as assessed by USS or Doppler, or confirmed by live birth.
Time Frame: After one or more FTET cycles, assessed at least 10 weeks after embryo transfer (up to 1 year)
Population: Participants enrolled in follow up study P05711 with vital pregnancy
Measure: Number; unit: Percentage of participants
Arm/Group | Corifollitropin Alfa 100 μg | recFSH 150 IU
Number analyzed (Participants) | 19 | 9
Percentage of participants | 0.0 | 0.0

4. Secondary Outcome: Percentage of Participants in Follow up Study With an Ecotopic Pregnancy
Description: An ectopic pregnancy is where the embryo implants outside the uterus. Ectopic pregnancies were calculated per total number of participants started in FTET.
Time Frame: After one or more FTET cycles, assessed at least 10 weeks after embryo transfer (up to 1 year)
Population: Participants enrolled in follow up study P05711
Measure: Number; unit: Percentage of participants
Arm/Group | Corifollitropin Alfa 100 μg | recFSH 150 IU
Number analyzed (Participants) | 77 | 25
Percentage of participants | 1.3 | 0.0

5. Secondary Outcome: Percentage of Participants in Follow up Study With a Clinical Pregnancy
Description: A clinical pregnancy is the presence of at least gestational sac or confirmed by live birth. Clinical pregnancies were calculated per attempt, meaning if any stage of in vitro fertilization (IVF) treatment was not achieved, zero values were imputed.
Time Frame: After one or more FTET cycles, assessed at least 10 weeks after embryo transfer (up to 1 year)
Population: Participants enrolled in follow up study P05711
Measure: Number; unit: Percentage of participants
Arm/Group | Corifollitropin Alfa 100 μg | recFSH 150 IU
Number analyzed (Participants) | 77 | 25
Percentage of participants | 28.6 | 40.0

6. Secondary Outcome: Percentage of Participants in Follow up Study With a Vital Pregnancy
Description: A vital pregnancy is the presence of at least one fetus with heart activity. Vital pregnancies were calculated per attempt, meaning if any stage of IVF treatment was not achieved, zero values were imputed.
Time Frame: After one or more FTET cycles, assessed at least 10 weeks after embryo transfer (up to 1 year)
Population: Participants enrolled in follow up study P05711
Measure: Number; unit: Percentage of participants
Arm/Group | Corifollitropin Alfa 100 μg | recFSH 150 IU
Number analyzed (Participants) | 77 | 25
Percentage of participants | 24.7 | 36.0

7. Secondary Outcome: Percentage of Participants With an Ongoing Pregnancy
Description: An ongoing pregnancy is the presence of at least one fetus with heart activity at least 10 weeks after embryo transfer or confirmed at live birth. Ongoing pregnancies were calculated per attempt, meaning if any stage of IVF treatment was not achieved, zero values were imputed.
Time Frame: After one or more FTET, assessed at least 10 weeks after embryo transfer or at live birth (up to 1 year)
Population: Participants enrolled in follow up study P05711
Measure: Number; unit: Percentage of participants
Arm/Group | Corifollitropin Alfa 100 μg | recFSH 150 IU
Number analyzed (Participants) | 77 | 25
Percentage of participants | 23.4 | 36.0

ADVERSE EVENTS:
Description: In Follow Up Study P05711, Serious Adverse Events (AEs) were not systematically monitored. Instead, any reported Serious AEs were unsolicited and non-systematically assessed. Other Adverse Events were not monitored and not collected.
Arm/Group | Corifollitropin Alfa 100 μg | recFSH 150 IU
Serious Adverse Events (participants affected / at risk) | 1/77 | 0/25
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Corifollitropin Alfa 100 μg (N=77) | recFSH 150 IU (N=25)
Cytogenetic abnormality (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor recognizes the right of the investigator(s) to publish, but all publications must be based on data validated and released by the Sponsor. Any such scientific paper, presentation, or other communication concerning the clinical trial described in this protocol will first be submitted to Sponsor, at least six weeks ahead of estimated publication or presentation, for written consent, which shall not be withheld unreasonably.